CLINICAL TRIAL: NCT01335984
Title: A Multi-center, Randomized, Parallel, Interventional, Open Label Trial to Compare the Blood Pressure-lowering Effect of Conventional Treatment and Smart Care Service in Hypertensive Patients Receiving Any Conventional Treatment
Brief Title: Effects of Telemonitoring and Telemedicine Service for Hypertensive Care
Acronym: Smart-HTN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Hee, Lee (Industry)
Collaborators: LG Electronics Inc. (Industry); Purdue University (Other)
Responsible Party: Sponsor-Investigator, Chang Hee, Lee, Chief Research Engineer, LG Electronics Inc.
Organization: LG Electronics Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SmartCare-HTN
Record Dates: First submitted 2011-03-31; First posted 2011-04-15 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Hypertension
Keywords: telemonitoring; usual care; telemedicine; telehealth; home care; Health Care Quality; Access; Evaluation
MeSH Terms: conditions — Hypertension | interventions — Telemedicine; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Telemonitoring group (Experimental): The subjects who are assigned in the Telemonitoring group should perform body composition measurement with self blood pressure measurement, and shall transmit the results to the Smart Care Serve via Smart Care PC. Telemonitoring group require site visit once per 2 months (8weeks)
  Interventions: Procedure: Telemonitoring
- Telemonitoring & Telemedicine group (Experimental): The subjects who are assigned in the Telemonitoring & Telemedicine group should perform body composition measurement with self blood pressure measurement, and shall transmit the results to the Smart Care Serve via Smart Care PC. Telemonitoring & Telemedicine group take remote medical treatment through video telephone instead of visiting study site.
  Interventions: Procedure: Telemonitoring & Telemedicine
- Control group (Other): The subjects who are assigned in the Control group require site visit once per 2 months (8weeks)
  Interventions: Other: control group

INTERVENTIONS:
Procedure: Telemonitoring — The subjects who are assigned in the Telemonitoring group will be provided Blood Pressure monitor, body composition analyzer, and remote monitoring device.
  The subjects who are assigned in the Telemonitoring group should visit the site once per every 2 months (8 weeks), and they should measure their blood pressure using a provided blood pressure monitor twice a day during study period (once after first morning urination and once before going to bed). After measurement of blood pressure and body composition, the subjects should make the transmission terminals of remote monitoring device situate near transmission terminal of Smart Care PC and transmit measured information through Smart Care PC into a centralized server of Smart Care Center.
  Other Names: Smartcare System : Telemonitoring
  Arms: Telemonitoring group
Procedure: Telemonitoring & Telemedicine — The subjects who are assigned in the Telemonitoring & Telemedicine group should perform the same remote monitoring procedures as the subjects in the Telemonitoring group.
  Since the remote visit substitute for a face to face visit, subjects should reserve the time for remote visit in each clinical trial center. A primary doctor or remote medical doctor should provide medical consultation to the subjects through videotelephony using the remote monitoring device and then issue electronic prescriptions.
  Other Names: Smartcare System : Telemonitoring & Telemedicine
  Arms: Telemonitoring & Telemedicine group
Other: control group — - The subjects who are assigned in the control group will be provided blood Pressure Monitor (Self BP measuring).
  The subjects who are assigned in the control group should perform the same blood pressure measurement (2 times a day) same as the test group during the study, and measured results should be recorded in a diary of self blood pressure measurement. In addition, the subjects should visit the site once per every two months (8 weeks).
  Other Names: Self-BP measuring
  Arms: Control group

SUMMARY:
This is a multi-centered, randomized, parallel group, interventional & open label clinical trial accessing efficacy of intervention effect by smart care system over existing treatment group for lowering blood pressure of hypertension patients taking anti-hypertension drug.

DETAILED DESCRIPTION:
1. Objectives : To evaluate superiority in blood pressure lowering effect of the Smart Care Service compared to the conventional treatment in hypertensive patients receiving any conventional antihypertensive medication
2. Test and control group

   * Control group : The subject group who is receiving any conventional treatment (hospital visit).
   * Test groups

   Conventional treatment + remote monitoring group:

   The subject group who is receiving the health care services using conventional treatment (hospital visit) and remote monitoring.

   Remote visit + remote monitoring group:

   The subject group who is receiving remote visit and remote monitoring using videotelephony
3. Target Subject: Hypertensive patients receiving any conventional antihypertensive medication

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients who are able to receive outpatient treatment from over 20 to under 70 years of age.- Over SBP 140mmHg without diabetes or renal failure
2. Patients who are taking more than one kind of any antihypertensive medications

   * Systolic blood pressure (SBP) ≥ 140mmHg in patient with diabetes mellitus and renal disease or
   * Systolic blood pressure (SBP) ≥ 130mmHg in patient without diabetes mellitus and renal disease
3. Patients who are able to understand the purpose of this trial and to read and write
4. Patients who are able to use Smart Care PC for this trial
5. Patients who participate voluntarily and sign the informed consent

Exclusion Criteria:

1. Patients with severe hypertension (mean of two seated SBP ≥200 mmHg) at screening visit blood pressure measurement.
2. Patients with secondary hypertension.
3. HbA1c>11%.
4. Patients are currently being hospitalized or planning to hospitalize due to hypertension.
5. Patients with severe renal disease (above 1.5 times the upper limit of normal serum creatinine levels).
6. Patients with any severe liver disease including cirrhosis (AST or ALT: above 3 times the upper limit of normal).
7. Patients who have been suffered cardiac infarction or severe coronary artery disease within 6 months, or with clinically significant congestive heart failure or heart valve defects.
8. Patients with phthisis, autoimmune disease or connective tissue disease.
9. Patients on medication therapies which may interfere with their blood pressure.
10. Patients with known history of allergic reaction or contraindication to angiotensin II antagonists.
11. Pregnant or lactating woman.
12. Patients with known history of alcoholism, mental illness, or drug dependency.
13. Patients who have participated in other study within 12 weeks prior to screening visit.
14. Any clinically significant medical condition including neurologic disease, gastrointestinal disease or malignant tumor, etc., which may affect the test results, or any other medical condition which in the opinion of the investigator makes the patients unsuitable for participation in the trial.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2011-01; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Clinic blood pressure | 24 weeks
  blood pressure value when hospital visiting
  * Clinic blood pressure
  * Changes in mean SBP(Systolic Blood Pressure) from baseline to 24 weeks visit

SECONDARY OUTCOMES:
Clinic blood pressure-Diastolic Blood Pressure(DBP) | 24 weeks
  Changes in mean Diastolic Blood Pressure(DBP) from baseline to 24 weeks visit
Percentage of subjects who achieved goal clinic blood pressure | 24 weeks
  Percentage of subjects who achieved blood pressure under 140/90mmHg at 24 weeks visit (under 130/80mmHg in subjects with diabetes mellitus and renal disease)
24 hours ABP(Ambulatory Blood Pressure) | 24 weeks
  * BP measured at baseline and after administration of antihypertensive drugs at 24 weeks
  * Mean values of 24 hours blood pressure (SBP / DBP) will be used for analysis
Percentage of subjects who achieved 24 hours ABP(Ambulatory Blood Pressure) goal | 24 weeks
  * Percentage of subjects who achieved average daytime BP of 24hrs ABPM under 135/85mmHg (under 130/80mmHg in subjects with diabetes mellitus and renal disease)
  * Average daytime BP will be calculated with average of each hourly mean from 07:00 to 22:59 of the Clock time
Self blood pressure measurement | 24 weeks
  Mean value of each week of self blood pressure measurement (Systolic/Diastolic) from baseline to 24 weeks
Medication compliance | 24 weeks
  * Patients diary will be recorded and medication compliance will be calculated by calculating the number of days administered antihypertensive drugs during the study
  * Drugs compliance = the number of days administered antihypertensive drugs / participated period in this study * 100%
Reduction of body mass index | 24 weeks
  Changes of Body Mass Index(BMI)
  - Body Mass Index(BMI)=Body weight (kg)/Height2(m) from baseline to 24 weeks
Assessment of patients' satisfaction | 24 weeks
  Only remote monitoring group and remote visit + remote monitoring group are applicable

CONTACTS AND LOCATIONS:
Overall Officials: Sungha Park, M.D., Principal Investigator — Yonsei University
Locations (3):
- South Korea (3):
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Medical Center, Daegu
  - Yonsei University Health System, Seoul